CLINICAL TRIAL: NCT00583453
Title: Perioperative Use of Celecoxib to Improve Pain Control in Patients Undergoing Tonsillectomy: a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Celecoxib as a Post-tonsillectomy Pain Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Douglas J Van Daele, Associate Professor of Otolaryngology-Head & Neck Surgery, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 200703765
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Tonsillitis
Keywords: Tonsillectomy; Analgesia; Pain measurement; Celecoxib
MeSH Terms: conditions — Tonsillitis; Agnosia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Celecoxib 200 mg tablets
  Interventions: Drug: Celecoxib
- B (Placebo Comparator): Placebo with same dosing schedule as the active comparator arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200 mg capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
  Other Names: Celebrex
  Arms: A
Drug: Placebo — Placebo capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
  Arms: B

SUMMARY:
The hypothesis is that celecoxib effectively reduces pain after a tonsillectomy and reduces post-operative narcotic use.

To test this hypothesis, the study is placebo controlled (sugar pill). Half of the participants will receive a sugar pill, half will not.

All participants will receive the standard post-operative pain medications.

We ask participants to log the amount of medications they use daily, and the amount of pain they have each day. It is hoped that celecoxib will reduce the amount of post-operative pain medication needed.

DETAILED DESCRIPTION:
Post-tonsillectomy pain is typically controlled through narcotic medications, such as Lortab elixir. Despite its standard use, this pain control is typically not as effective as a non-steroidal anti-inflammatory medication (NSAID). The problem with using NSAIDs for post-tonsillectomy operative pain is the significant increased risk of rebleeding.

Celecoxib is an NSAID that is a COX-2 inhibitor; the drug is designed to act as an NSAID without the increased risk of rebleeding or hemorrhage.

This study is a double blind, randomized study; neither the study participant or the study investigator knows if the participant is receiving celecoxib or a placebo (sugar pill). The blinded list is maintained by the research pharmacists and can be unblinded when needed (such as in an emergency).

Participants begin taking the study medication the night before surgery and continue through 10 days post-operative. Participants are asked to complete a journal that catalogs the amount of standard post-operative medications taken, the amount of pain experienced, and any other comments.

Participants are contacted by phone at 5 and 10 days post-op.

Study participation ends at the standard 3-week post-operative check-up.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Indication for tonsillectomy (patients undergoing a tonsillectomy as a portion of additional surgical procedures will not be included)
* Have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of bleeding disorders
* History of liver or kidney dysfunction
* History of allergy to sulfa containing medications
* History of lactose intolerance
* History of asthma, urticaria, or allergic-type reactions to aspirin or NSAIDs
* Women who are currently pregnant, nursing, or trying to conceive
* History of allergy or intolerance to acetaminophen or hydrocodone
* History of allergy to any COX-2 inhibitor, including celecoxib or rofecoxib.
* PT, PTT, hemoglobin, or hematocrit values that are outside of institutional limits.
* History of cardiovascular disease
* Patients currently taking celecoxib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas VanDaele, MD, Principal Investigator — Department of Otolaryngology-Head & Neck Surgery
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded through clinicaltrials.gov data tables

REFERENCES:
- [Result] Van Daele DJ, Bodeker KL, Trask DK. Celecoxib Versus Placebo in Tonsillectomy: A Prospective, Randomized, Double-Blind Placebo-Controlled Trial. Ann Otol Rhinol Laryngol. 2016 Oct;125(10):785-800. doi: 10.1177/0003489416654707. Epub 2016 Jun 29. PMID 27357971

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib as Experimerimental Intervention: Celecoxib 200 mg tablets
  Celecoxib: Celecoxib 200 mg capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
- Placebo Control, Active Comparator: Placebo with same dosing schedule as the active comparator arm
  Placebo: Placebo capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
Period: Overall Study
Arm/Group | Celecoxib as Experimerimental Intervention | Placebo Control, Active Comparator
Started | 9 | 8
Completed | 9 | 6
Not Completed | 0 | 2
Not completed — discontinued intervention | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib 200 mg Tablets: Celecoxib 200 mg tablets
  Celecoxib: Celecoxib 200 mg capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
- Placebo With Same Dosing Schedule as the Active Comparator Arm: Placebo with same dosing schedule as the active comparator arm
  Placebo: Placebo capsule
  1. capsule the night before surgery
  2. capsules the morning of surgery
  1 capsule the night of surgery
  1 capsule twice daily for 10 days immediately after the surgery
- Total: Total of all reporting groups
Arm/Group | Celecoxib 200 mg Tablets | Placebo With Same Dosing Schedule as the Active Comparator Arm | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (4.1) | 25.0 (3.3) | 25.0 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Pain Score
Description: Pain score as reported by participant, measured on a 10 point scale, where 0 = none and 10 = unbearable, collected once daily.
Time Frame: day of procedure through post-operative day 10
Measure: Mean (Standard Error); unit: pain score (units on a scale)
Arm/Group | Celecoxib 200 mg Tablets | Placebo With Same Dosing Schedule as the Active Comparator Arm
Number analyzed (Participants) | 9 | 6
pain score (units on a scale)
  Maximum pain, day 1 | 5.0 (0.6) | 6.0 (0.7)
  maximum pain, averaged across days 2 to 4 | 5.1 (0.6) | 6.0 (0.7)
  maximum pain, averaged across days 5 to 7 | 4.4 (0.6) | 5.9 (0.7)
  maximum pain, averaged across days 8 to 10 | 3.6 (0.6) | 4.0 (0.7)
  Average pain, day 1 | 6.1 (1.0) | 7.3 (0.8)
  Average pain, averaged across days 2 to 4 | 6.2 (0.9) | 7.6 (0.8)
  Average pain, averaged across days 5 to 7 | 6.1 (0.9) | 7.4 (0.8)
  Average pain, averaged across days 8 to 10 | 4.9 (0.9) | 5.7 (0.8)
  Pain with drinking, day 1 | 5.7 (0.9) | 6.7 (0.8)
  Pain with drinking, averaged across days 2 to 4 | 5.4 (0.8) | 6.6 (0.7)
  Pain with drinking, averaged across days 5 to 7 | 4.9 (0.8) | 5.9 (0.7)
  Pain with drinking, averaged across days 8 to 10 | 3.9 (0.8) | 4.1 (0.7)
  Activity, day 1 | 2.8 (0.9) | 4.5 (1.0)
Statistical Analysis 1: Comparison: Celecoxib 200 mg Tablets vs Placebo With Same Dosing Schedule as the Active Comparator Arm; Test type: Superiority or Other; p = .674, Wilcoxon (Mann-Whitney) — Treatment x day interaction

2. Secondary Outcome: Self-reported Activity Level
Description: Activity level, reported by participant utilizing a 10-point ordinal scale (0 = no activity, 10 = return to normal activities). Activity level was measured was collected once daily.
Time Frame: From operative day through 10 days post-operative
Measure: Mean (Standard Error); unit: Activity score (units on a scale)
Arm/Group | Celecoxib as Experimerimental Intervention | Placebo Control, Active Comparator
Number analyzed (Participants) | 9 | 6
Activity score (units on a scale)
  Day 1 | 2.8 (0.9) | 4.5 (1.0)
  Average, days 2 to 4 | 3.1 (0.7) | 4.1 (0.9)
  Average, days 5 to 7 | 5.4 (0.7) | 3.7 (0.9)
  Average, days 8 to 10 | 7.4 (0.7) | 5.7 (0.9)
Statistical Analysis 1: Comparison: Celecoxib as Experimerimental Intervention vs Placebo Control, Active Comparator; Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney) — Treatment x day interaction reported as 0.018

3. Secondary Outcome: Acetaminophen Equivalent Use
Description: Participant reported acetaminophen use and its equivalent. Medication use was collected from reported participant journals.
Time Frame: From operative day through 10 days post-operative
Measure: Mean (Standard Error); unit: mg
Arm/Group | Celecoxib as Experimerimental Intervention | Placebo Control, Active Comparator
Number analyzed (Participants) | 9 | 6
mg
  Day 1 | 2074 (407) | 3006 (498)
  Average, days 2 to 4 | 2245 (356) | 2934 (436)
  Average, days 5 to 7 | 2028 (356) | 3610 (436)
  Average, days 8 to 10 | 1418 (356) | 2483 (436)
Statistical Analysis 1: Comparison: Celecoxib as Experimerimental Intervention vs Placebo Control, Active Comparator; Test type: Superiority or Other; p = .214, Wilcoxon (Mann-Whitney) — Treatment x day interaction = 0.214

4. Secondary Outcome: Incidence of Post-operative Hemorrhage
Description: The incidence of post-operative hemorrhage, defined as post-operative bleeding requiring medical intervention or hospitalization during the 10 day post-operative follow-up period.
Time Frame: From operative day through 10 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib 200 mg Tablets | Placebo With Same Dosing Schedule as the Active Comparator Arm
Number analyzed (Participants) | 9 | 6
Participants | 0 | 0

5. Secondary Outcome: Total Morphine Equivalent
Description: Participant reported mophine equivalent use
Time Frame: From operative day through 10 days post-operative
Measure: Mean (Standard Error); unit: mg
Arm/Group | Celecoxib as Experimerimental Intervention | Placebo Control, Active Comparator
Number analyzed (Participants) | 9 | 6
mg
  Day 1 | 28.9 (11.6) | 55.0 (14.2)
  Average, days 2 to 4 | 30.4 (9.6) | 72.4 (11.7)
  Average, days 5 to 7 | 27.8 (9.6) | 69.7 (11.7)
  Average, days 8 to 10 | 13.2 (9.6) | 38.3 (11.7)
Statistical Analysis 1: Comparison: Celecoxib as Experimerimental Intervention vs Placebo Control, Active Comparator; Test type: Superiority or Other; p = 0.036, Wilcoxon (Mann-Whitney) — treatment x day interaction P = 0.036 Treatment main effect (average day 1 to 10) P = 0.003

ADVERSE EVENTS:
Time Frame: 3 weeks postoperatively
Arm/Group | Celecoxib as Experimerimental Intervention | Placebo Control, Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 1/9 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib as Experimerimental Intervention (N=9) | Placebo Control, Active Comparator (N=6)
Vomiting, grade 1 (Gastrointestinal disorders) | 1 (5) | 2 (2) — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Dehydration, grade 2 (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — A disorder characterized by excessive loss of water from the body. It is usually caused by severe diarrhea, vomiting or lack of adequate fluid intake. Grade 2: I.V. fluids indicated for less than 24 hours
Dysphagia, grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1) — A disorder characterized by difficulty in swallowing. Grade 2 = symptomatic and altered eating / swallowing

LIMITATIONS AND CAVEATS:
Small sample size Disproportionately female population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No